CLINICAL TRIAL: NCT01025661
Title: Effects of Chiropractic Care on Pain and Function in Patients With Hip Osteoarthritis Waiting for Arthroplasty - a Controlled Clinical Pilot Trial
Brief Title: Effects of Chiropractic Care in Patients With Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scandinavian College of Chiropractic (Other)
Collaborators: Karolinska Institutet (Other); Stockholm South General Hospital (Other)
Responsible Party: Gordana Gedin, Head Principal, Scandinavian College of Chiropractic
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2007/7900-31/3
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-12

CONDITIONS: Hip Osteoarthritis
Keywords: chiropractic; hip osteoarthritis; hip arthroplasty; pain; activities of daily living.
MeSH Terms: conditions — Osteoarthritis, Hip; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Waiting list control (No Intervention): The waiting list controls did not receive any intervention during the study period.
  Interventions: Other: Chiropractic care

INTERVENTIONS:
Other: Chiropractic care — Clinical examinations and treatments were performed at the outpatient clinic. The patients were assessed and treated by research assistants and the clinical care was supervised by state registered chiropractors. The choice of therapy and modality was pragmatic and based on the analysis of different functions such as mobility, tenderness, muscle tension and tone, and each patient's relative symptoms. Chiropractic care included high-velocity and low-amplitude techniques, soft-tissue or myofascial techniques, and arthrokinematic stabilizing exercises or a combination of these. Patients were treated in 1-2 sessions per week during the trial.

SUMMARY:
The purpose of the study is to explore the short term effects of chiropractic care on pain and function in patients with hip osteoarthritis.

DETAILED DESCRIPTION:
Research over the last years have reported a scarce of trails investigating chiropractic treatment of lower extremities. Osteoarthritis, also called joint failure, is a common rheumatic joint disease often affecting the hipjoint, contributing to pain, decreased mobility and loss of function. Individuals with osteoarthritis can also be affected in many other ways, e.g. economically, socially and emotionally.

Chiropractic care may be considered as a complement to the conventional allopathic treatment of hip osteoarthritis. Joint manipulation is a well-established treatment technique to restore optimal joint function of the locomotor system. The aim of the study is to explore the effects of chiropractic vs. continued conventional care (waiting list controls) on pain and function during a three week trail period among patients with hip osteoarthritis waiting for arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* waiting for first time unilateral arthroplasty on the affected side

Exclusion Criteria:

* documented osteoporosis, current pathology such as malignancy, infection, cardiovascular disease, stroke and femoral fractures on affected side

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)

PRIMARY OUTCOMES:
The 100mm Visual Analogue Scale (VAS) | Baseline and follow up after three weeks

SECONDARY OUTCOMES:
The five sub-scales of the Hip disability and Osteoarthritis Outcome Score (HOOS), i.e. pain, other symptoms, function in daily living (ADL), function in sport and recreation (sport/rec) and hip related Quality of life (QOL) | Baseline and follow up after three weeks

CONTACTS AND LOCATIONS:
Overall Officials: P M Thorman et al, RC, Principal Investigator — Skandinavian College Of Chiropractic
Locations (1):
- Scandinavian College of Chiropractic, Solna, Stockholm County, Sweden